CLINICAL TRIAL: NCT04263506
Title: A Vignette-based Randomized Controlled Trial to Evaluate the Impact of Supervisor's Role on Research Practices of Doctoral Students Facing Dilemma Situations
Brief Title: A Vignette-based Randomized Controlled Trial to Evaluate the Impact of Supervisor's Role on Research Practices of Doctoral Students
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: ISB-014
Record Dates: First submitted 2020-02-07; First posted 2020-02-10 (Actual); Last update posted 2020-02-10 (Actual); Status verified 2020-01

CONDITIONS: The Study Focus on no Specific Condition

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Vignette with supervisor's opinion (Experimental): Participants in this arm will receive vignettes with an additional sentence describing supervisor's opinion (i.e. supervisor does not oppose to detrimental research practice)
  Interventions: Other: Vignette with emphasis on supervisor's opinion
- Vignette without supervisor's opinion (Active Comparator): Participants in this arm will receive vignettes without an additional sentence describing supervisor's opinion.
  Interventions: Other: Vignette with emphasis on supervisor's opinion

INTERVENTIONS:
Other: Vignette with emphasis on supervisor's opinion — A vignette describing a dilemma situation for a researcher (e.g. adding an honorary author) with or without the description of supervisor's advice that does not oppose to detrimental research practice (i.e. the supervisor is fine with whatever the PhD student decides in the dilemma).

SUMMARY:
This study aims to evaluate the influence of supervisors on PhD students' research practice (i.e., an environment where there is a lack of opposition to detrimental research practice from the supervisor)

DETAILED DESCRIPTION:
PhD students are the next generation of researchers and will present the field in the future. However, several environmental factors might influence their research practice. In this study, we will evaluate the influence of supervisors on PhD students' research practice (an environment where there is a lack of opposition to detrimental research practice from the supervisor).

Objective: To evaluate the influence of supervisors on PhD students' research practice

Design: A randomized controlled trial

1. Intervention: Participants will be shown two case vignettes describing dilemma situations in research reported with and without the role of the supervisor.
2. Participants: The participants will be PhD students in all biomedical disciplines.
3. Sample size will be 300 participants
4. Primary outcome: In each vignette, participants will have to indicate which solution they prefer on a semantic differential scale, rated from - 5 to -1 (preference for solution A) and from 1 to 5 (preference for solution B). Participants will be forced to make a choice between the 2 solutions. The primary outcome will be the mean preference score.
5. This study is approved by ethics review regulations by INSERM (CEEI-IRB): IRB00003888

ELIGIBILITY:
Inclusion Criteria:

* PhD students in biomedical sciences

Exclusion Criteria:

* NA

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 300 (Estimated)
Dates: Start 2020-03-01 (Estimated); Primary Completion 2020-12-01 (Estimated); Study Completion 2020-12-01 (Estimated)

PRIMARY OUTCOMES:
Mean preference score | Immediate assessment
  In each vignette, we will ask participants, what would you do if you are in the place of the character in the vignette? Participants will have to indicate which solution they prefer on a semantic differential scale, rated from - 5 to -1 (preference for solution A) and from 1 to 5 (preference for solution B). We will calculate the mean preference score

SECONDARY OUTCOMES:
Proportion of students who chose the detrimental research practice | Immediate assessment
  Proportion of students who made choices rated from -5 to -1

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Nguyen VT, Sharp MK, Superchi C, Baron G, Glonti K, Blanco D, Olsen M, Vo Tat TT, Olarte Parra C, Neveol A, Hren D, Ravaud P, Boutron I. Biomedical doctoral students' research practices when facing dilemmas: two vignette-based randomized control trials. Sci Rep. 2023 Sep 29;13(1):16371. doi: 10.1038/s41598-023-42121-1. PMID 37773192